CLINICAL TRIAL: NCT01100645
Title: Efficacy and Safety of the Herbal Medicine Sominex ® (Passiflora Incarnata L., Valeriana Officinalis L. and Crataegus Oxyacantha L.), Manufactured by the Laboratory EMS S / A in Patients With Psychophysiological Insomnia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clínica Pesquisa e Desenvolvimento Ltda.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VCPEMS0210; Version 2
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-04

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Test (Experimental): Sominex ® (Passiflora incarnata L. 50 mg, Valeriana officinalis L. 40 mg and Crataegus oxyacantha L. 30 mg)
  Interventions: Drug: Sominex
- Placebo (Placebo Comparator): Excipient
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sominex — Passiflora incarnata L.50 mg Valeriana officinalis L.40 mg Crataegus oxyacantha L.30 mg
  Arms: Test
Drug: Placebo — Excipient
  Arms: Placebo

SUMMARY:
The main objective of this study is to evaluate the clinical efficacy of the drug Sominex (Valeriana officinalis L., 40 mg, 30 mg Crataegus oxyacantha L. and Passiflora incarnata L. 50 mg) manufactured by the Laboratory EMS S / A, compared to placebo in improving sleep efficiency, based on the response of the sleep quality questionnaire (MSQ) and polysomnographic parameters described below:

* Latency to onset of sleep;
* Total time of sleep;
* Rapid eye movement (REM) sleep latency;
* Duration of REM sleep

DETAILED DESCRIPTION:
Verify the effectiveness of the drug Sominex compared to placebo based on the improvement of the following parameters measured by the following validated scales:

* Anxiety;
* Daytime sleepiness; Will also be assessed secondary to drug safety testing for the occurrence, type, frequency and intensity of adverse events during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who agree and sign the informed consent form (ICF);
2. Adult patients, aged ≥ 18 years and ≤ 65 years, male or female;
3. Patients who agree to perform all study procedures;
4. Patients diagnosed with psychophysiological insomnia;
5. Patients who present in the application of sleep questionnaire result ≥ 25 and ≤ 30 points;
6. Patients presenting in polysomnography change in any of the polysomnographic parameters than the normal range.

Exclusion Criteria:

1. Having participated in any experimental study or have ingested any drug trial within 12 months prior to the start of the study;
2. Be in use or have used other medications that interfere with the regular response of the drug at least 04 weeks prior to the start of the study, as benzodiazeínicos, antidepressants with sedative, sedatives, antihistamines and other herbal medicines;
3. Being in treating or have been treated with alternative methods that interfere with the drug response to at least 04 weeks prior to the start of the study, such as behavioral therapies and relaxation techniques, such as yoga, massage, etc.;
4. Be patient with sensitivity to an association of herbal medicines;
5. Present history of alcohol abuse, drugs or medicines;
6. Pregnant or nursing women;
7. Owning a history of liver disease or renal impairment and / or thyroid dysfunction;
8. Patients with a history of restless sleep: nocturnal myoclonus or restless legs syndrome;
9. Patients with a history of snoring or bruxism exaggerated;
10. Diseases that affect sleep, causing pain or immobilization of the patient in bed;
11. Patients who have extensive work or working in night shifts totally or partially nocturnal;
12. Patients in whom polysomnography demonstrating non-characteristic changes in sleep disturbances of psychophysiological origin as narcolepsy, hipopinéia syndrome, upper airway hypersensitivity syndrome of periodic limb movements, sleepwalking, among others;
13. Physical or psychological disorders that might interfere with the analysis of data such as neurosis, depression, muscle atrophy, and / or staying the medical criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-01 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Improvement in sleep efficiency | 28 days of treatment.
  Quality of Sleep Questionnaire and the polysomnographic parameters:
  * Latency to onset of sleep;
  * Total time of sleep;
  * REM sleep latency;
  * Duration of REM sleep;

SECONDARY OUTCOMES:
Improvement of the values obtained by the answers of the questionnaires obtained during the treatment | 28 days of treatment.
  Scale Hamilton Anxiety (HAM-A); Daytime Sleepiness Scale Epworth; Journal of Sleep

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clinica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil